CLINICAL TRIAL: NCT03556761
Title: Furosemide for Accelerated Recovery of Blood Pressure Postpartum
Acronym: ForBP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Lisa Levine, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 829444
Record Dates: First submitted 2018-06-01; First posted 2018-06-14 (Actual); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Hypertension, Pregnancy-Induced
Keywords: Furosemide; Postpartum; Hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension | interventions — Furosemide

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, placebo control design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study medication (furosemide) and placebo will be stored at room temperature at the University of Pennsylvania research pharmacy. Pharmacy will be responsible for labeling and randomizing the medications.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral furosemide (Experimental): Oral furosemide 20 mg/day for a total of 5 consecutive doses.
  Interventions: Drug: Oral furosemide
- Placebo Oral Tablet (Placebo Comparator): Placebo once per day for a total of 5 consecutive doses.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Oral furosemide — Furosemide (Lasix), 20 milligram, PO, PO, daily
  Arms: Oral furosemide
Drug: Placebo Oral Tablet — Placebo, PO, daily
  Arms: Placebo Oral Tablet

SUMMARY:
A randomized, double-blind, placebo-controlled single center investigation of furosemide's effect on postpartum blood pressure control in pregnancies affected by hypertensive disorders of pregnancy

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy are recognized causes of significant maternal/fetal morbidity and mortality, accounting for approximately 18% of maternal deaths worldwide. While significant research has been done on the evaluation and management of hypertension during pregnancy, studies of postpartum hypertension (PPHTN) are usually limited by their retrospective design and focus on inpatients in the immediate postpartum period (2-6 days), or patients who were readmitted due to complications related to hypertension. Few studies have investigated the incidence and proper management of hypertension in the postpartum period. Furthermore, in the United Kingdom, a review of maternal deaths determined that 10% were related to hypertensive disorders in pregnancy (HDP) in the postpartum period. Postpartum hypertension is also the cause of approximately 27% of readmissions to the hospital. These studies clearly show that PPHTN is associated with significant morbidity and that it is important to develop interventions that can reduce its effects.

In patients with HDP, postpartum blood pressure has been shown to decrease in the first 48 hours postpartum only to then increase in days 3-6 postpartum. This phenomenon is thought to be secondary to large fluid shifts, both secondary from fluid retention during the pregnant state as well as from fluids given intrapartum. Furthermore, large volumes of sodium are also mobilized into the intravascular compartment at this time. Given the latter, furosemide, a loop diuretic that mobilizes sodium and fluid excretion has been posed as a method to prevent severe range blood pressures and their associated maternal morbidity in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive disorder of pregnancy diagnosed antepartum or intrapartum
* Gestational hypertension
* Pre-eclampsia with or without severe features
* Superimposed pre-eclampsia with or without severe features
* New diagnosis of HDP within 24 hours from delivery
* Postpartum, delivery ≥ 20 weeks estimated gestational age
* Age ≥18 years old

Exclusion Criteria:

* History of allergic reaction to furosemide
* High risk comorbidities for which treatment may be indicated or contraindicated: class C or higher diabetes mellitus, chronic kidney disease or baseline creatinine >1.2, cardiac disorders including cardiomyopathy, congenital heart disease, angina or coronary heart disease, rheumatic disease (lupus), sickle cell disease
* Baseline labs with K <3
* Use of furosemide or other diuretics antepartum or intrapartum
* Use of ototoxic agents including aminoglycosides (ie, Gentamicin for >1 dose), cephalosporins (ie Ancef >1 dose),
* Patient unstable for protocol per investigator's judgement

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 384 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2020-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Levine, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopes Perdigao J, Lewey J, Hirshberg A, Koelper N, Srinivas SK, Elovitz MA, Levine LD. Furosemide for Accelerated Recovery of Blood Pressure Postpartum in women with a hypertensive disorder of pregnancy: A Randomized Controlled Trial. Hypertension. 2021 May 5;77(5):1517-1524. doi: 10.1161/HYPERTENSIONAHA.120.16133. Epub 2021 Feb 8. PMID 33550824

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Furosemide | Placebo Oral Tablet
Started | 192 | 192
Completed | 168 | 163
Not Completed | 24 | 29

BASELINE CHARACTERISTICS:
Groups:
- Oral Furosemide: Oral tablet of furosemide 20 mg once daily for a total of 5 consecutive doses.
- Placebo Oral Tablet: Oral tablet of placebo once daily for a total of 5 consecutive doses.
- Total: Total of all reporting groups
Arm/Group | Oral Furosemide | Placebo Oral Tablet | Total
Number analyzed (Participants) | 192 | 192 | 384
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [22 to 32] | 27 [23 to 33] | 27 [22 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192 | 192 | 384
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 151 | 138 | 289
  White | 30 | 47 | 77
  Other | 11 | 7 | 18
Hypertensive Disorders of Pregnancy (HDP) [Count of Participants; unit: Participants]
  Non-severe | 128 | 133 | 261
  Severe | 64 | 59 | 123
Gestational age at delivery [Median (Inter-Quartile Range); unit: weeks] | 38.6 [37.3 to 39.7] | 38.4 [37.3 to 39.7] | 38.5 [37.3 to 39.7]
Cesarean delivery [Number; unit: participants] | 55 | 38 | 93

OUTCOME MEASURES:

1. Primary Outcome: Persistently Elevated Blood Pressures 7 Days Postpartum
Description: To compare the rate of persistently elevated blood pressures (>140/90) in women that receive a five day furosemide course compared to those that receive placebo.
Time Frame: 0-7 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Furosemide | Placebo Oral Tablet
Number analyzed (Participants) | 168 | 163
Participants | 10 | 23
Statistical Analysis 1: Comparison: Oral Furosemide vs Placebo Oral Tablet; Test type: Superiority; p = 0.03, Regression, Linear; Risk Ratio (RR) = 0.40, 95% CI 2-sided [0.20 to 0.81]

2. Primary Outcome: Time to Resolution
Description: To compare the time (days) required to achieve a resolution of elevated blood pressure, adjusted for mode of delivery.
Time Frame: 0-14 days postpartum
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Oral Furosemide | Placebo Oral Tablet
Number analyzed (Participants) | 168 | 163
days | 10 [6.25 to 12.5] | 10.5 [6.5 to 12.5]
Statistical Analysis 1: Comparison: Oral Furosemide vs Placebo Oral Tablet; Test type: Superiority; p = 0.12, Regression, Cox; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.95 to 1.51]

3. Secondary Outcome: Postpartum Readmission
Description: Number of subjects with one or more readmission/ER visit that were hypertension related
Time Frame: 0-6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Furosemide | Placebo Oral Tablet
Number analyzed (Participants) | 168 | 163
Participants | 9 | 16
Statistical Analysis 1: Comparison: Oral Furosemide vs Placebo Oral Tablet; Test type: Superiority; p = 0.14, Chi-squared; Risk Ratio (RR) = 0.55, 95% CI 2-sided [0.25 to 1.21]

4. Secondary Outcome: Number of Subjects Who Had Severe Hypertension Postpartum
Description: Number of women who had severe hypertension (systolic blood pressure>160 millimeters of mercury or diastolic blood pressure>110 millimeters of mercury) postpartum
Time Frame: 0-6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Furosemide | Placebo Oral Tablet
Number analyzed (Participants) | 168 | 163
Participants | 81 | 86
Statistical Analysis 1: Comparison: Oral Furosemide vs Placebo Oral Tablet; Test type: Superiority; p = 0.36, Chi-squared; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.64 to 1.18]

5. Secondary Outcome: Postpartum Length of Stay
Description: Number of days postpartum participants stayed in the hospital
Time Frame: 0-6 weeks postpartum
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Oral Furosemide | Placebo Oral Tablet
Number analyzed (Participants) | 168 | 163
Days | 2 [2 to 3] | 2 [2 to 2]
Statistical Analysis 1: Comparison: Oral Furosemide vs Placebo Oral Tablet; Test type: Superiority; p = 0.76, Regression, Linear; Risk Ratio (RR) = 0.02, 95% CI 2-sided [-0.09 to .13]

6. Secondary Outcome: Subjects With Complications During Hospitalization
Description: Subjects with complications during hospitalization related to hypertensive disorders of pregnancy.
Time Frame: 0-6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Furosemide | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 192
Participants | 3 | 1
Statistical Analysis 1: Comparison: Oral Furosemide vs Placebo Oral Tablet; Test type: Superiority; p = 0.62, Fisher Exact

7. Secondary Outcome: Number of Subjects Experiencing One or More Adverse Effects
Description: Number of subjects experiencing one or more adverse effects secondary to furosemide
Time Frame: 0-6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Furosemide | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 192
Participants | 0 | 1
Statistical Analysis 1: Comparison: Oral Furosemide vs Placebo Oral Tablet; Test type: Superiority; Risk Ratio (RR) = 3, 95% CI 2-sided [0.32 to 28.59]

8. Secondary Outcome: Number of Subjects That Required for Additional Antihypertensives
Description: Number of subjects that required additional hypertensive medication after discharge
Time Frame: 0 to 6 weeks post-partum
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Furosemide | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 192
Participants | 25 | 39
Statistical Analysis 1: Comparison: Oral Furosemide vs Placebo Oral Tablet; Test type: Superiority; p = 0.03, Chi-squared; Risk Ratio (RR) = 0.61, 95% CI 2-sided [0.39 to 0.96]

ADVERSE EVENTS:
Time Frame: Over 6 weeks postpartum
Arm/Group | Oral Furosemide | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/192 | 0/192
Serious Adverse Events (participants affected / at risk) | 0/192 | 0/192
Other Adverse Events (participants affected / at risk) | 3/192 | 1/192
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Furosemide (N=192) | Placebo Oral Tablet (N=192)
Pulmonary edema (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1) — Pulmonary edema

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT03556761/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT03556761/ICF_001.pdf